CLINICAL TRIAL: NCT04022655
Title: Predictors of Mortality in Patients With Autoimmune Diseases Admitted to the Intensive Care Unit - Retrospective Analysis at a Single Tertiary Care Center
Brief Title: Predictors of Mortality in Patients With Autoimmune Diseases Admitted to the Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Göttingen (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Peter Korsten, Attending Physician, Head of the Rheumatology Clinical Trials Unit, Prinicipal Investigator, University of Göttingen
Other Study IDs: 4/8/19
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Vasculitis; Systemic Lupus Erythematosus; Myositis
Keywords: Intensive Care Unit; Mortality; Autoimmune Diseases
MeSH Terms: conditions — Vasculitis; Lupus Erythematosus, Systemic; Myositis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ANCA-associated Vasculitis: Patients with ANCA-associated vasculitis admitted to the ICU
  Interventions: Other: ICU Care

INTERVENTIONS:
Other: ICU Care — No intervention

SUMMARY:
Autoimmune diseases, such as systemic lupus erythematosus, rheumatoid arthritis, myositis, or anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis, may affect multiple organ systems. Occasionally, patients deteriorate acutely requiring advanced care in an intensive care unit (ICU). In an ICU setting, mortality is estimated with scoring systems, such as APACHE or SAPSII. Since there are limited data available on their use in autoimmune diseases, with the current study, we aim to assess the usefulness of these ICU scores and analyze predictors of mortality in this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU at the University Medical Center Göttingen

Exclusion Criteria:

* Patients with incomplete or missing data

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with systemic autoimmune diseases admitted to the ICU at the University Medical Center Göttingen
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | From date of admission to the ICU until the date of death from any cause assessed up to 52 weeks

SECONDARY OUTCOMES:
Risk of renal replacement therapy | From date of admission to the ICU until the date of event assessed up to 52 weeks
Need for catecholamines | From date of admission to the ICU until the date of event assessed up to 52 weeks
Need for ventilation | From date of admission to the ICU until the date of event assessed up to 52 weeks
Need for cardiopulmonary resuscitation | From date of admission to the ICU until the date of event assessed up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Korsten, MD, Principal Investigator — University Medical Center Göttingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No